CLINICAL TRIAL: NCT01331629
Title: Impact of Art Therapy on Fatigue and Quality of Life of Patients Treated With Adjuvant Radiotherapy for Breast Cancer
Acronym: ART-THERAPIE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ART-THERAPIE
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; fatigue; quality of life; art-therapie; adjuvant radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ART-THERAPIE (Experimental): supported in art therapy with other supportive care available in the facility
  Interventions: Other: ART-THERAPIE
- standard group (No Intervention): standard care (supportive care available in each facility)

INTERVENTIONS:
Other: ART-THERAPIE — 8 sessions of art therapy during radiotherapy
  Arms: ART-THERAPIE

SUMMARY:
The purpose of this study is to compare intervention by Art-therapy to standard care in patients treated with adjuvant radiotherapy for breast cancer and evaluate the fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer surgery (invasive or in situ) by conservative surgery
* Age ≥ 18 years
* Indication of adjuvant radiotherapy
* Adjuvant chemotherapy allowed
* Agreeing to participate in a clinical study
* Able to participate in a clinical trial

Exclusion Criteria:

* Metastatic Breast Cancer
* Personal history of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
evaluate persistent fatigue | up to 12 months after radiotherapy
  Estimate the decrease in the proportion of patients with persistent fatigue after one month of radiotherapy in patients receiving an approach from art therapy as a complement to standard care compared to those with care standard alone.
  Evaluated by auto-questionnary

SECONDARY OUTCOMES:
Evaluate the quality of life patients. | up to 12 months after radiotherapy
  Evaluate the quality of life patients (by auto-questionnary)
Assess the impact of the condition of patients on the reactions, depression and anxiety of relatives Assess the impact of the condition of patients on the reactions, depression and anxiety of relatives | up to 12 months after radiotherapy
  Assess the impact of the condition of patients on the reactions, depression and anxiety of relatives (by auto-questionnary)
Evaluate the fatigue away from the treatment (at 6 months and 1 year) of patients | 6 months and 12 months after treatment
  Evaluate the fatigue away from the treatment (at 6 months and 1 year) of patients (by auto-questionnary)
Evaluate the anxiety of patients | up 12 months after radiotherapy
  Evaluate the anxiety of patients (by auto-questionnary)
evaluate the depression of patients | up 12 months after study
  evaluate the depression of patients (by auto-questionnary)
Evaluate the quality of life away from the treatment (at 6 months and 1 year) of patients | 6 months and 1 year after treatment
  Evaluate the quality of life away from the treatment (at 6 months and 1 year) of patients (by auto-questionnary)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre François BACLESSE, Caen, Calvados
  - CHU, Grenoble, Isère
  - Centre Oscar LAMBRET, Lille, Nord
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - Centre Antoine LACASSAGNE, Nice
  - Institut Jean Godinot, Reims